CLINICAL TRIAL: NCT02620176
Title: The Effect of Transcutaneous Vagal Nerve Stimulation on Reducing Oesophageal Pain Hypersensitivity in Healthy Volunteers
Brief Title: The Effect of Transcutaneous Vagal Nerve Stimulation on Reducing Oesophageal Pain Hypersensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wingate Institute of Neurogastroenterology (Other)
Responsible Party: Principal Investigator, Adam Farmer, PhD MRCP, Wingate Institute of Neurogastroenterology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Farmer-2
Record Dates: First submitted 2014-12-15; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous vagal nerve stimulation (Experimental): Active vagal nerve stimulation to the left auricular branch of the vagus nerve.
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Sham vagal nerve stimulation (Placebo Comparator): Placebo vagal nerve stimulation stimulation. The stimulator is attached to the left ear, but rotated 180 degrees, so that it is not stimulating the auricular branch of the vagal nerve.
  Interventions: Device: Transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — Trans-auricular vagal nerve stimulation
  Other Names: NEMOS

SUMMARY:
We are evaluating the role of transcutaneous electrical vagal nerve stimulation in the prevention of oesophageal pain hypersensitivity using a validated human model in healthy volunteers.

DETAILED DESCRIPTION:
Chronic oesophageal pain is a symptomatic feature of disorders such as erosive oesophagitis, non-erosive reflux disease and non-cardiac chest pain. Patients often display heightened sensitivity to intra-oesophageal stimuli, which is referred to as oesophageal pain hypersensitivity. However, the experience of oesophageal pain is highly individual with a multitude of factors proposed to account for this variability. Amongst the physiological factors is the autonomic nervous system (ANS). The ANS has been postulated to play a pivotal role in the modulation of pain through its multiple interactions with pain processing. The ANS has two broadly antithetic branches, the parasympathetic nervous system (PNS) and the sympathetic nervous system (SNS). The primary neural substrate of the PNS is the vagus nerve. The vagus nerve is increasingly considered to play an integral role in modulating oesophageal pain. Electrical vagal nerve stimulation (VNS) was first used in humans in 1988 and is an efficacious treatment for drug resistant epilepsy. Traditional VNS is undertaken in a procedure where a bipolar helical electrode is placed around the cervical vagal nerve, which is connected to a pulse generator placed in subcutaneous pocket in the chest, not dissimilar to a cardiac pacemaker. However, this method of VNS necessitates surgical implantation with its attendant risks and complications. Recently, an external transcutaneous VNS (t-VNS) system, consisting of an earplug-like electrode to interface with the concha of the outer ear and a handheld battery-powered electrical stimulator, has become commercially available (NEMOS system). The auricular branch of the vagus nerve innervates the concha of the ear and is located directly under the skin, making it a suitable target for transcutaneous stimulation. t-VNS has been demonstrated to be safe, well tolerated and have a high degree of user-friendliness. A preliminary study has reported that t-VNS reduces sensitivity to heat pain in healthy volunteers. Furthermore, recent studies have demonstrated that t-VNS patterns of cerebral activation, as determined by functional magnetic resonance imaging, were similar to those evoked by traditional VNS. Thus, VNS per se represents an attractive proposition for investigating the role of the PNS in oesophageal pain and t-VNS specifically, a viable, safe and acceptable technology for achieving this. The pivotal experiments evaluating the analgesic role of VNS in the development of acid induced oesophageal pain hypersensitivity have not been conducted. Using the aforementioned model of oesophageal pain hypersensitivity, we seek to determine the analgesic effect of t-VNS.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide Informed written consent
* Healthy volunteers aged 18-65, who have no medical history

Exclusion Criteria:

* Any inclusion criteria not met
* Subjects unable to provide informed consent.
* Subjects with any systemic disease or medications that may influence the autonomic nervous system (e.g. beta-agonists or Parkinson's disease).
* Pregnant females to prevent any confounding effects on pregnancy related nausea.
* Subjects who suffer from reflux disease
* Subject who take any medication, including over the counter preparations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Sensitisation to electrical stimuli in the proximal oesophagus following a distal oesophageal acid infusion in comparison to baseline | 90 minutes post acid infusion
  Pain tolerance thresholds to electrical stimulation in the proximal oesophagus decrease following a distal oesophageal acid infusion due to central sensitisation and are defined as a reduction of >6mA in thresholds. Prevention of sensitisation will be defined as this threshold not being met.

SECONDARY OUTCOMES:
Sensitisation to electrical stimuli in the proximal oesophagus following a distal oesophageal acid infusion in comparison to baseline | 30 minutes post acid infusion
  Pain tolerance thresholds to electrical stimulation in the proximal oesophagus decrease following a distal oesophageal acid infusion due to central sensitisation and are defined as a reduction of >6mA in thresholds. Prevention of sensitisation will be defined as this threshold not being met.
Sensitisation to electrical stimuli in the proximal oesophagus following a distal oesophageal acid infusion in comparison to baseline | 60 minutes post acid infusion
  Pain tolerance thresholds to electrical stimulation in the proximal oesophagus decrease following a distal oesophageal acid infusion due to central sensitisation and are defined as a reduction of >6mA in thresholds. Prevention of sensitisation will be defined as this threshold not being met.
Effect of vagal nerve stimulation on cardiac vagal tone during stimulation in comparison to baseline | 30 minutes
  The effect of vagal stimulation on the validated parameter of cardiac vagal tone
Effect of vagal nerve stimulation on cardiac sympathetic index during stimulation in comparison to baseline | 30 minutes
  The effect of vagal stimulation on the validated parameter of cardiac sympathetic index.

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute of Neurogastroenterology, London, London, United Kingdom

REFERENCES:
- [Background] Botha C, Farmer AD, Nilsson M, Brock C, Gavrila AD, Drewes AM, Knowles CH, Aziz Q. Preliminary report: modulation of parasympathetic nervous system tone influences oesophageal pain hypersensitivity. Gut. 2015 Apr;64(4):611-7. doi: 10.1136/gutjnl-2013-306698. Epub 2014 May 28. PMID 24870622
- See also: Description: Vagal nerve stimulator information — http://www.cerbomed.com